CLINICAL TRIAL: NCT07291843
Title: The Effects of Vibration Therapy and Instrument-Assisted Soft Tissue Mobilization on Pain, Range of Motion, Functionality, Joint Position Sense, and Quality of Life in Individuals With Subacromial Impingement Syndrome
Brief Title: Vibration Therapy and IASTM in Subacromial Impingement Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emre DANSUK (Other)
Responsible Party: Sponsor-Investigator, Emre DANSUK, Principal Investigator, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7891
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Impingement Syndrome; Impingement Shoulder; Shoulder Pain
Keywords: Subacromial Impingement Syndrome; Shoulder Pain; Instrument-Assisted Soft Tissue Mobilization (IASTM); Vibration Therapy; Physiotherapy
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: This study uses a three-arm parallel-group randomized controlled design in which participants diagnosed with subacromial impingement syndrome are randomly assigned to one of three intervention groups: (1) Vibration Therapy combined with Conventional Physiotherapy, (2) Instrument-Assisted Soft Tissue Mobilization (IASTM) combined with Conventional Physiotherapy, or (3) Conventional Physiotherapy alone. All groups receive interventions three times per week for four weeks. Outcomes are compared between groups to determine the additional effects of vibration therapy and IASTM beyond standard physiotherapy.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy (Active Comparator): All participants will receive a total of 12 sessions of conventional therapy and exercise, administered three days per week for four weeks. The conventional therapy program will include 8 minutes of ultrasound, 30 minutes of TENS (Transcutaneous Electrical Nerve Stimulation), and 15 minutes of cryotherapy.
  The exercise program will consist of passive stretching performed by the physiotherapist, as well as supervised exercises including Codman pendulum exercises, wand-assisted exercises, finger ladder exercises, and strengthening exercises tailored to the patient's condition. All exercises will be applied progressively based on the participant's tolerance and clinical status.
  Interventions: Other: Conventional physiotherapy
- Vibration Therapy Group (Experimental): Participants in this group will receive vibration therapy in addition to conventional physiotherapy methods. The vibration application (33 Hz) will be administered using a percussion massage device (Compex Fixx 2.0) to the M. Deltoideus, M. Supraspinatus, M. Infraspinatus, and M. Teres Minor muscles. The treatment will be applied along the origin-to-insertion line of each muscle for 3 minutes per muscle.
  The device will be moved in a straight longitudinal path along the muscle fibers, progressing from proximal to distal and then returning to the proximal segment. Each stroke will last approximately five seconds. Vibration therapy will be applied using the soft-head attachment of the percussion device.
  The vibration intervention will be carried out three times per week for a total of four weeks.
  Interventions: Device: Percussion massage therapy device; Other: Conventional physiotherapy
- IASTM Group (Experimental): In the IASTM group, participants will receive instrument-assisted soft tissue mobilization three days per week for four weeks, for a total of 12 sessions, following the conventional physiotherapy treatment. The technique will be applied with the participant in a supine position to the anterior muscle groups, including the subscapularis, anterior deltoid, pectoralis major, pectoralis minor, and biceps brachii muscles. The participant will then be placed in a prone position to treat the posterior muscle groups, including the upper trapezius, supraspinatus, infraspinatus, teres major, teres minor, and posterior deltoid muscles. Each muscle group will receive treatment at a 45-degree angle using sweep and brush techniques, consisting of 20 seconds of parallel strokes and 20 seconds of perpendicular strokes.
  Interventions: Device: Instrument-assisted soft tissue mobilization device; Other: Conventional physiotherapy

INTERVENTIONS:
Device: Percussion massage therapy device — Vibration therapy was applied using a handheld percussion massage gun (Compex Fixx 2.0) delivering vibration at 33 Hz with a soft-head attachment. The device was moved longitudinally along the deltoid and rotator cuff muscles (supraspinatus, infraspinatus, teres minor) in a proximal-to-distal direction. Each muscle was treated for approximately 3 minutes per session. The intervention was delivered three times per week for four weeks.
  Arms: Vibration Therapy Group
Device: Instrument-assisted soft tissue mobilization device — Instrument-assisted soft tissue mobilization was performed using specially designed stainless-steel tools applied at a 45-degree angle to the anterior and posterior shoulder muscles. Sweep and brush techniques were used, consisting of approximately 20 seconds of parallel strokes and 20 seconds of perpendicular strokes per muscle group. The intervention was administered three times per week for four weeks following the conventional physiotherapy session.
  Arms: IASTM Group
Other: Conventional physiotherapy — Conventional physiotherapy consisting of 8 minutes of therapeutic ultrasound, 30 minutes of TENS, 15 minutes of cryotherapy, and a supervised exercise program including passive stretching, Codman pendulum exercises, wand exercises, finger ladder exercises, and progressive strengthening. The program is delivered three times per week for four weeks.

SUMMARY:
This randomized controlled clinical study aims to investigate the effects of vibration therapy and instrument-assisted soft tissue mobilization (IASTM), when added to conventional physiotherapy, on pain, range of motion, proprioception, functional status, and quality of life in individuals diagnosed with subacromial impingement syndrome (SAIS). SAIS is one of the most common causes of shoulder pain and is frequently associated with impaired scapular kinematics, rotator cuff dysfunction, soft tissue tightness, and decreased shoulder mobility.

A total of 48 participants aged 40-60 years with MRI-confirmed SAIS will be randomly assigned into three groups: (1) Vibration Therapy + Conventional Physiotherapy, (2) IASTM + Conventional Physiotherapy, and (3) Conventional Physiotherapy (Control). All interventions will be administered three times per week for four weeks. Outcomes include pain intensity (VAS), shoulder range of motion (Goniometer Pro app), proprioception at 60° of flexion and abduction, functional status (DASH), and quality of life (RC-QoL).

The study aims to determine whether adding vibration therapy or IASTM to standard physiotherapy provides additional short-term benefits in reducing pain, improving joint mobility, enhancing proprioceptive acuity, and increasing functional capacity in individuals with subacromial impingement syndrome.

DETAILED DESCRIPTION:
Subacromial impingement syndrome (SAIS) is one of the most frequently encountered musculoskeletal disorders, affecting approximately 20-30% of the general population and representing a major cause of shoulder pain. SAIS has been associated with altered scapular kinematics, rotator cuff muscle imbalance, soft-tissue tightness, postural abnormalities, and impaired neuromuscular control. Conventional physiotherapy-including therapeutic exercises, stretching, electrotherapy modalities, and manual techniques-is commonly used in clinical practice. However, evidence suggests that combining manual or soft-tissue-based interventions with standard physiotherapy may yield more effective improvements in pain, mobility, and shoulder function.

Instrument-assisted soft tissue mobilization (IASTM) is a manual therapy technique that uses ergonomically designed stainless steel tools to provide controlled mechanical stimulation to soft tissues. IASTM has recently gained attention due to its ability to increase soft-tissue extensibility, promote myofascial release, and enhance joint range of motion. Similarly, vibration-based interventions-including percussion massage therapy-have been shown to improve circulation, decrease pain, reduce muscle stiffness, and enhance mobility through mechanical oscillation and stimulation of sensory receptors. Despite their growing popularity, limited evidence exists regarding the direct comparison of vibration therapy and IASTM in individuals with SAIS.

This randomized controlled trial aims to evaluate whether adding vibration therapy or IASTM to conventional physiotherapy provides superior outcomes compared with conventional physiotherapy alone. A total of 48 adults aged 40-60 years with MRI-confirmed SAIS will be randomly allocated into three groups: (1) Vibration Therapy + Conventional Physiotherapy, (2) IASTM + Conventional Physiotherapy, and (3) Conventional Physiotherapy (Control). All interventions will be delivered three times per week for four weeks. Vibration therapy will be applied using a percussion massage device (33 Hz) to the deltoid and rotator cuff muscles along the origin-to-insertion path. IASTM will be applied using standardized sweep and brush techniques at a 45° angle to both anterior and posterior shoulder muscle groups. The control group will receive conventional physiotherapy consisting of ultrasound, TENS, cryotherapy, passive stretching, Codman exercises, wand exercises, finger ladder exercises, and progressive strengthening, supervised by a physiotherapist.

Outcome measures include pain intensity (VAS), shoulder range of motion measured with the Goniometer Pro mobile application, proprioception assessed at 60° flexion and abduction, functional disability evaluated using the DASH questionnaire, and shoulder-related quality of life measured with the RC-QoL scale. Assessments will be conducted at baseline and after the 4-week intervention period.

This study seeks to contribute to the current literature by directly comparing two frequently used soft-tissue interventions-vibration therapy and IASTM-within the SAIS population. The findings are expected to inform clinicians about the potential added benefits of combining these modalities with conventional physiotherapy to optimize pain reduction, functional improvement, and neuromuscular outcomes in individuals with subacromial impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with subacromial impingement syndrome confirmed by MRI
* Men and women between 40 and 60 years of age
* Presence of symptoms for more than one month

Exclusion Criteria:

* History of surgery on the affected arm
* Presence of an open wound on the arm
* Existing infection
* Inflammatory joint disease
* Shoulder osteoarthritis
* Presence of rheumatic disease
* Malignant or benign tumors
* Inability to tolerate vibration therapy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Joint Position Sense (Proprioception) | 4 week
  Joint position sense will be assessed using the Becure Extremity ROM system. Proprioception will be evaluated at 60 degrees of shoulder flexion and shoulder abduction. While standing, each participant will first be asked to lift their arm with eyes open and memorize the arm position at 60 degrees. Then, with eyes closed, the participant will be instructed to raise the arm to the same position previously reached with eyes open. The shoulder angle will be measured while the eyes are closed.
  The difference between the angles recorded with eyes open and eyes closed will be considered the joint position error. This procedure will be performed for both shoulder flexion and abduction at 60 degrees.

SECONDARY OUTCOMES:
Pain Assessment (Visual Analog Scale - VAS) | 4 week
  The Visual Analog Scale (VAS) is a commonly used method for assessing pain intensity. Participants will be asked to mark the level of pain they perceive on a 100-mm horizontal line. The left end of the line represents no pain, while the right end represents the worst imaginable pain. The distance measured from the left end to the participant's mark will be recorded as the pain score.
Range of motion (ROM) | 4 week
  Shoulder range of motion (ROM) of the participants will be measured using the Becure Extremity ROM system. Flexion and abduction will be assessed within a 0-180° range, while internal and external rotation will be evaluated within a 0-90° range.
Functionality (Disabilities of the Arm, Shoulder and Hand Questionnaire - DASH) | 4 week
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is used to assess physical disability and functional status in individuals with upper extremity disorders. The questionnaire consists of three subsections. The first section includes 30 items designed to evaluate the patient's functional level and symptoms. Of these 30 items, 21 assess the individual's ability to perform daily activities, 5 evaluate symptoms (pain, activity-related pain, tingling, weakness, and stiffness), and the remaining 4 address social functioning, work, sleep, and confidence in performing activities.
  The optional Work Module consists of 4 questions and is used to evaluate the patient's ability to perform work-related tasks. Each item is rated on a 5-point Likert scale (1 = no difficulty, 2 = mild difficulty, 3 = moderate difficulty, 4 = severe difficulty, 5 = unable to perform). Higher scores indicate greater disability and more severe functional limitation.
Quality of Life (Rotator Cuff Quality of Life Questionnaire - RC-QoL) | 4 week
  The scale is a condition-specific assessment tool designed to measure quality of life in individuals with rotator cuff pathologies.
  The questionnaire consists of 34 items grouped under five domains, including physical symptoms, work-related activities, activities of daily living, social functioning, and emotional well-being. Each item is scored on a scale from 0 to 100, where "0" indicates severe pain and "100" indicates no pain. Higher scores reflect better quality of life.
  The total score is calculated by summing the scores of all completed items, dividing the sum by the number of answered questions, and then converting the result into a percentage value.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Dansuk, PhD, Principal Investigator — Medipol University
Locations (1):
- Emre Dansuk, Istanbul, Beykoz, Turkey (Türkiye)